CLINICAL TRIAL: NCT06547450
Title: Study of the Cost-efficacy and Acceptability of the Unified Protocol for Treatment of Emotional Disorders in Brief Groups in Primary Care Services in Spain (PU-AP)
Brief Title: Unified Protocol for Treatment of Emotional Disorders in Brief Groups in Primary Care Services in Spain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Jorge Javier Osma López, Principal Investigator, Instituto de Investigación Sanitaria Aragón
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2023-151473OB-100
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-08

CONDITIONS: Emotional Disorder; Anxiety Disorders; Depressive Disorder
Keywords: Emotional Disorder; Unified Protocol; Primary Care; Transdiagnostic approach; Group format; Brief format
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: All consecutive patients with emotional disorders attending any of the collaborating centers will be asked to participate in the present study. Once inclusion criteria are met, each patient will be randomly assigned to one of the two experimental groups: the 8-session UP group or the 5-session UP group. Randomization will be performed by a researcher unrelated to the study using a computer-generated sequence (Randomizer). Randomization will be stratified according to the severity of the primary measures of depression and anxiety, using the recommended cutoff in the manuals. Stratification will be made to ensure a comparable proportion of severely depressed and anxious individuals in each group. For each subgroup (i.e., severe or less severe depression and/or anxiety), participants will be randomly assigned to the 8-session UP group or the 5-session UP group.
Who Masked: Outcomes Assessor
Masking Description: Patients (participants) will know the treatment they have been assigned to. Healthcare professionals and researchers will know the condition each patient has been assigned to (mandatory to provide a given type of intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5-session UP condition (Experimental): In both conditions, the contents of the UP manual were worked following the 2nd edition of the UP manual (Barlow et al., 2018). In the 5-session version, modules 1 (Motivation for change and commitment to treatment) and 8 (Achievement, maintenance, and relapse prevention) were removed and modules 6 and 7 (interoceptive and emotional exposure) were combined. The sessions were group sessions, 2 hours long and weekly.
  Interventions: Behavioral: 5-session UP condition
- 8-session UP condition (Active Comparator): In both conditions, the contents of the UP manual were worked following the 2nd edition of the UP manual (Barlow et al., 2018). In the 8-session UP condition, each of the original 8 treatment modules was worked on per week. The sessions were group sessions, 2 hours long and weekly.
  Interventions: Behavioral: 8-session UP condition

INTERVENTIONS:
Behavioral: 5-session UP condition — Unified Protocol (UP) for transdiagnostic treatment of EDs in 5-session
  Arms: 5-session UP condition
Behavioral: 8-session UP condition — Unified Protocol (UP) for transdiagnostic treatment of EDs in 8-session
  Arms: 8-session UP condition

SUMMARY:
The aim of this project is to contribute to the improvement of psychological care received in primary care (PC), through the study of the cost-effectiveness and acceptability of the Unified Protocol for the treatment of emotional disorders in brief groups in primary care services in Spain (PU-AP) for the treatment of emotional disorders (EDs), the most prevalent in our society. To do so, a pilot study will be carried out, and, subsequently, a randomized clinical trial to study the efficacy, cost-effectiveness and acceptability of the Unified Protocol for the transdiagnostic treatment of EDs, applied in 5 or 8 group sessions. Finally, the researchers will analyze whether there are specific patient profiles that will benefit more from one or the other condition. The results will contribute to the personalization of the psychological treatment of users with EDs attending PC in the Spanish public health system.

DETAILED DESCRIPTION:
Emotional disorders (EDs;including anxiety disorders, unipolar mood disorders, and related disorders) are the most prevalent mental disorders in the general population. In Spain, anxiety disorders and mood disorders affect approximately two million (4.1%) and two and half million (5.2%) individuals, respectively. As a result of their prevalence in the society, EDs have become an alarming health problem due to their associate costs. These disorders have a direct cost of 22.000 million euros (500 euros per capita and year). The total expense of these disorders entails 2.2% of the Gross Domestic Product in Spain.

In recent years, several alternatives have been proposed to address this situation, one of them being an increase in the number of clinical psychologists in our national health system (NHS) and, especially, their incorporation into primary care (PC) services.

It is considered that the incorporation of psychology in PC will help to reduce referral to specialized care because it will be possible to carry out a more exhaustive screening and determine which cases do not require psychological treatment, which cases should be referred to other health care resources and which cases can be treated in PC, usually mild-moderate TE. Another alternative to mitigate the excessive demand for care, regardless of the level of care, is the use of group psychological interventions, a cost-effective format for systems with limited resources such as our NHS.

Transdiagnostic interventions, like the Unified Protocol for the Treatment of EDs (UP), in brief group format, has emerged as a viable option for treating EDs in PC services.

The aim of the present study is to analyze the efficacy, cost-effectiveness and acceptability of the Unified Protocol for the transdiagnostic treatment of EDs, applied in 5 or 8 group sessions.

Furthermore, it will try to find out which characteristics of the participants (e.g., gender, clinical diagnoses, transdiagnostic dimensions affected, symptom severity) predict a better outcome (e.g., clinical improvement and quality of life) as a function of the sessions received. Thus, in the future, it will be possible to offer the optimal number of sessions according to specific profiles (personalization of treatments).

ELIGIBILITY:
Inclusion Criteria:

* Have at least one EDs diagnosis (anxiety, depressive, obsessive-compulsive, trauma and somatic disorders) from the ADIS-5 interview
* Have a score between 0 and 5 severity (mild-moderate) on the diagnoses on the CSR of the ADIS-5
* Be able to attend all assessment and treatment sessions
* Individuals on pharmacological treatment will be asked to maintain the dosage for the duration of the study, unless there is a medical contraindication

Exclusion Criteria:

* Absence of clinical diagnosis
* Presenting a diagnosis of EDs with a severity score on diagnoses between 6 and 8 on the ADIS-5 CSR (severe) or a clinical condition requiring specialized mental health intervention such as presence of severe mental disorder (e.g., personality disorder, bipolar disorder, or schizophrenia), suicide risk at the time of assessment, or substance use in the past three months
* Who have received 8 or more sessions of CBT (during the past five years) with techniques such as cognitive flexibility or exposure
* Who are receiving psychological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS-V) | Enrollment and Up to 6 months
  Diagnostic interview
  Diagnostic interview
Overall Depression Severity and Impairment Scale (ODSIS) | Up to 6 months
  Consist of five items that evaluate the frequency and the intensity of depressive symptoms and their interference with the person's work or school life and social life. The total score range from 0 to 20 and responses use a 5-point Likert scale ranging from 0 to 4.
Overall Anxiety Severity and Impairment Scale (OASIS) | Up to 6 months
  The scale presents five items. These items are related with the frequency and intensity of anxiety symptoms and their interference with the person's work or school life and with social life. All items are rated on a 5-point Likert scale ranging from 0 (I didn't feel anxious) to 4 (Constant anxiety).
Health-related quality of life (EuroQol-5D) | Up to 6 months
  Evaluation through 5 items of quality of life. For this study, the visual analog scale (EQ-VAS) was used, using a score from 0 to 100 (0 = worst imaginable state of health; 100 = best imaginable state of health).
Difficulties in Emotion Regulation Scale (DERS) | Up to 6 months
  Consists of 36-item of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation

SECONDARY OUTCOMES:
The Multidimensional Emotional Disorder Inventory (MEDI) | Up to 6 months
  A self-report measure that includes only 49 items and enables to quickly assess the main transdiagnostic dimensions of Emotional disorders: neurotic temperament (MEDI_NT), positive temperament (MEDI_PT), depressed mood (MEDI_DM), autonomic arousal (MEDI_AA), somatic anxiety (MEDI_SOM), intrusive cognitions (MEDI_IC), social concerns (MEDI_SOC), traumatic re-experiencing (MEDI_TRM), and avoidance (MEDI_AVD). It uses a 9-point Likert-type response scale (0 = Does not characterize me; 8 = Totally characterizes me).
Five Facet Mindfulness Questionnaire (FFMQ) | Up to 6 months
  Is a 39-item questionnaire that measures five facets of mindfulness. responses use a 5-point Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true)
Working Alliance Inventory-Short (WAI-S) | Up to 6 months
  Evaluate the therapeutic or working alliance through 12 items grouped in three dimensions, called task (1, 2, 10 and 12), links (3, 5, 7 and 9) and objectives (4, 6, 8 and 11) measured through a Likert-type scale with scores ranging from 1 = Never to 7 = Always.
Maladjustment Scale (MI) | Up to 6 months
  Evaluates interference in different vital areas through six items with a 6-point Likert-type response scale (0 = Not at all; 5 = Extremely).
Positive and negative affect scale | Up to 6 months
  Evaluates the dimensions of positive and negative affect, through 20 items and is rated on a 5-point scale from 1 (not at all) to 5 (very much).
Adaptation of Client Satisfaction Questionnaire [CSQ-8] | Up to 6 months
  An adaptation of 13 items that measures quality of the intervention and its components, discomfort experienced during treatment through the following 7 questions with a 4-point Likert-type response scale (0 = nothing; 3 =very much): 1) How would you rate the quality of the treatment program you received?; 2) Did you find the kind of psychological intervention you were looking for?; 3) If a friend or family member needed similar help, would you recommend our treatment program?; 4) Has the content you have learned helped you cope more effectively with your problems?; 5) Overall, how satisfied are you with the treatment program you received?; 6) To what extent has this treatment program caused you discomfort?; 7) If you had to seek help again, would you choose a group treatment program?
Quality-adjusted Life Years (QALYs) | Up to 6 months
  Measure of disease burden, including both the quality and the quantity of life lived. It is used in economic evaluation to assess the value of medical interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Osma, Ph.D, Principal Investigator — Instituto de Investigación Sanitaria de Aragón, Universidad de Zaragoza
Locations (1):
- Centro de Salud Carinyena, Hospital Universitario de La Plana, Villarreal, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Under request

REFERENCES:
- [Background] Barlow DH, Harris BA, Eustis EH, Farchione TJ. The unified protocol for transdiagnostic treatment of emotional disorders. World Psychiatry. 2020 Jun;19(2):245-246. doi: 10.1002/wps.20748. No abstract available. PMID 32394551
- [Derived] Peris-Baquero O, Fadrique-Jimenez A, Prieto-Rollan I, Camacho-Guerrero L, Martinez-Lluesma S, Osma J. Brief Versions of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Spanish Primary Care Service: Results of a Feasibility Pilot Study. J Clin Psychol. 2025 Nov;81(11):1103-1117. doi: 10.1002/jclp.70016. Epub 2025 Jul 16. PMID 40667676
- See also: Related Info — http://www.iisaragon.es/grupos-de-investigacion/neurociencia-salud-mental-y-organos-de-los-sentidos/giis082-investigacion-en-personalidad-emocion-y-salud-ipes/
- See also: Related Info — http://www.alianzaeditorial.es/libro/manuales/aplicaciones-del-protocolo-unificado-para-el-tratamiento-transdiagnostico-de-la-disregulacion-emocional-jorge-osma-9788491817260/
- See also: Related Info — http://www.alianzaeditorial.es/libro/manuales/protocolo-unificado-para-el-tratamiento-transdiagnostico-de-los-trastornos-emocionales-manual-del-terapeuta-david-h-barlow-9788491814795/
- See also: Related Info — http://www.alianzaeditorial.es/libro/manuales/protocolo-unificado-para-el-tratamiento-transdiagnostico-de-los-trastornos-emocionales-manual-del-paciente-david-h-barlow-9788491814818/
- See also: IPES web (Investigation group) — http://ipes-group.com/